CLINICAL TRIAL: NCT06931938
Title: Awake PROne Positioning in PatientS With Acute Hypoxemic Respiratory Failure in Germany - A Randomized Controlled Study
Brief Title: Awake Prone Positioning in Spontaneous Breathing Patients With Acute Hypoxic Respiratory Failure Due to Pneumonia
Acronym: PROSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Charite University, Berlin, Germany (Other); Asklepios Klinikum Harburg (Unknown); University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Stefan Kluge, MD, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-101424-BO-ff
Record Dates: First submitted 2025-04-09; First posted 2025-04-17 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Acute Hypoxemic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Awake prone positioning (Active Comparator): The clinical intervention in the Intervention Group is Awake Prone Positioning, a standard therapy in intensive care units worldwide in ARDS care. The intervention should not be started later than 24 hours after randomization. An earlier start, as soon as possible, after randomization is strongly recommended. In patients in the intervention group standard Awake Prone Positioning for at least 10 hours/day for a length of 72 hours should be applied. The reach the targeted 10 hours / day (per 24 hours), it is strongly recommended to use blocks of a longer time period (e.g. multiple 3-5 hours blocks) within the 24h period to reach the anticipated APP goal. It is recommended that the APP therapy within the targeted intervention for 10 hours/day (per 24 h period) is not interrupted for more than 2 hours till reaching the goal of 10 hours/day (per 24h). It is further strongly recommended that one APP session should last at least 3 hours. (...) For more information please see the protocol.
  Interventions: Other: Awake Prone Positioning
- Standard supine/semi-recumbent positioning (No Intervention): Patients randomized to the control arm will receive standard positioning at the discretion of the treating team but excluding APP. Control group patients will remain in their natural choice of position, which is anticipated to favour a supine, semi-recumbent position. The use of awake prone positioning as a so-called rescue intervention is discouraged in the control group and recorded as a protocol violation.
  If patients have to be tracheal intubated and mechanically ventilated treatment should follow current ARDS guidelines. This includes PP in patients with mild to severe ARDS if PaO2/FiO2 is below 150 mmHg.

INTERVENTIONS:
Other: Awake Prone Positioning — The clinical intervention in the Intervention Group is Awake Prone Positioning, a standard therapy in intensive care units worldwide in ARDS care. The intervention should not be started later than 24 hours after randomization. An earlier start, as soon as possible, after randomization is strongly recommended. In patients in the intervention group standard Awake Prone Positioning for at least 10 hours/day for a length of 72 hours should be applied. The reach the targeted 10 hours / day (per 24 hours), it is strongly recommended to use blocks of a longer time period (e.g. multiple 3-5 hours blocks) within the 24h period to reach the anticipated APP goal. It is recommended that the APP therapy within the targeted intervention for 10 hours/day (per 24 h period) is not interrupted for more than 2 hours till reaching the goal of 10 hours / day (per 24 h). It is further strongly recommended that one APP session should last at least 3 hours. (...) For more information please see the protol.
  Arms: Awake prone positioning

SUMMARY:
Prone positioning has shown beneficial effects in intubated patients with severe respiratory failure and positive effects in awake patients with COVID-19 pneumonia. Conclusive evidence for patients with AHRF without COVID-19 is still missing. The investigators hypothesis that awake prone position in patients with AHRF is superior to standard supine/semi-recumbent position in terms of reducing the rate of tracheal intubation and/or all-cause death within 28 days after randomization.

DETAILED DESCRIPTION:
Prone positioning has shown beneficial effects in intubated patients with severe respiratory failure and positive effects in awake patients with COVID-19 pneumonia. Since the pandemic the rate of awake prone positioning has increased and became a standard medical therapy in ICUs worldwide. Conclusive evidence for patients with AHRF without COVID-19 is still missing. The investigators hypothesize that awake prone position in patients with AHRF is superior to standard supine/semi-recumbent position in terms of reducing the rate of tracheal intubation and/or all-cause death within 28 days after randomization. Furthermore, the investigators aim to assess safety and tolerability of awake prone positioning in patients with acute hypoxic respiratory failure due to pneumonia on the ICU.

ELIGIBILITY:
Inclusion Criteria:

* The focus of this trial is to treat patients with respiratory failure. The inclusion criteria are selected accordingly. Patients meeting all of the criteria listed below will be included in the study:

  * Patients in the intensive care unit
  * High possibility of Pneumonia (community-acquired pneumonia or hospital-acquired pneumo-nia) either diagnosed by chest x-ray or computed tomography or clinically diagnosed at least with one of the following signs

    * Appearance of purulent secretions or changes in characteristics (color, odor, quantity, consistency)
    * Cough or dyspnea or tachypnea
    * Evocative auscultation
  * Presence of acute hypoxemic respiratory failure (PaO2/FIO2 ≤ 300 mmHg or SpO2/FiO2 ≤ 315)

Exclusion Criteria:

* Patients are excluded from the study if any of the following criteria are met at screening or before ran-domization, a detailed list is shown in the study manual:

  * Age below 18
  * Pregnant woman
  * Patient is unlikely/unable to awake prone positioning, or to be compliant as indicated by the treating team
  * Prolonged need (≥ 4 days) for HFNO, NIV or CPAP before study inclusion
  * Urgent need for endotracheal intubation
  * Invasive Mechanical Ventilation
  * Shock

    o Defined as need for vasopressor ≥ 0.4 mcg/kg/min to maintain a mean blood pressure of ≥ 65 mmHg or systolic blood pressure ≥ 90 mmHg
  * Participation in another clinical interventional trial in the last 3 months
  * Previous Participation in the PROSA Trial
  * Long-term oxygenation therapy (LTOT) or continuous positive airway pressure (CPAP) therapy before hospital admission
  * Treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Tracheal intubation and/or all-cause death | 28 days
  Tracheal intubation and/or all-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Kluge, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual anonymized patient data underlying the results of the publication
Supporting Information: Study Protocol, ICF, CSR
Time Frame: up to 36 Months after publication of results
Access Criteria: Upon resonable request

DOCUMENTS (1):
  • Study Protocol (2024-12-28): https://cdn.clinicaltrials.gov/large-docs/38/NCT06931938/Prot_000.pdf